CLINICAL TRIAL: NCT01013870
Title: The Mission Connect Mild TBI Translational Research Consortium's Integrated Clinical Protocol
Brief Title: Mission Connect Mild Traumatic Brain Injury (TBI) Integrated Clinical Protocol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to recruit adequate numbers of subjects
Sponsor: Baylor College of Medicine (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Claudia Sue Robertson, Professor, Department of Neurosurgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-08-2-0132
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Results first posted 2016-11-17 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Traumatic Brain Injury; Post-traumatic Stress Disorder
Keywords: mild traumatic brain injury; post-concussion syndrome; acute stress disorder; post-traumatic stress disorder; atorvastatin
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Brain Concussion; Post-Concussion Syndrome; Stress Disorders, Traumatic, Acute | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MTBI subjects randomized to drug (Experimental): Of 200 MTBI subjects enrolled, 1:1 randomization will be used to assign half (i.e 100) to the treatment arm of the phase II drug trial of atorvastatin. These subjects will receive a daily weight-based dose of atorvastatin 1mg/kg (up to 80 mg) for seven days and started within 24 hours of MTBI, and their outcome will be compared with the group of subjects receiving a placebo.
  NOTE: The 100 Orthopedic Injury subjects recruited for and participating in the Observational studies are not included in the Medication study portion of this protocol.
  Interventions: Drug: Atorvastatin
- MTBI subjects randomized to placebo (Placebo Comparator): Of 200 MTBI subjects enrolled, 1:1 randomization will be used to assign half (i.e 100) to the placebo arm of the phase II drug trial of atorvastatin. These subjects will receive a daily dose of an inert preparation, visually indistinguishable from the active agent. They will take this preparation for seven days, started within 24 hours of MTBI, and their outcome will be compared with the group of subjects receiving active drug.
  NOTE: The 100 Orthopedic Injury subjects recruited for and participating in the Observational studies are not included in the Medication study portion of this protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — In this Phase II randomized clinical trial of 200 MTBI subjects to evaluate atorvastatin as a neuroprotective agent, subjects will receive either active drug or placebo (1:1 randomization) for 7 days, starting within 24 hours of the brain injury. The dosage for subjects in the treatment group will be weight-based at 1mg/kgm, up to 80 mg, which will be the maximal dose. Subjects will be monitored at 3-4 days after injury by phone, then with follow-up visits at 1 week, 1 month, 3 months.
  Other Names: Lipitor®
  Arms: MTBI subjects randomized to drug
Drug: Placebo — In this Phase II randomized clinical trial of 200 MTBI subjects to evaluate atorvastatin as a neuroprotective agent, subjects will receive either active drug or placebo (1:1 randomization) for 7 days, starting within 24 hours of the brain injury. For the placebo group, subjects will take a daily dose of an inert preparation, visually indistinguishable from the active agent. They will take this preparation for seven days, started within 24 hours of MTBI, and their outcome will be compared with the group of subjects receiving active drug. Subjects will be monitored at 3-4 days after injury by phone, then with follow-up visits at 1 week, 1 month, 3 months.
  Arms: MTBI subjects randomized to placebo

SUMMARY:
The purpose of this study is to improve the ability to diagnose problems after mild traumatic brain injury (MTBI) and to test a drug that may improve the outcome from these injuries. Of the more than 1.5 million people who experience a traumatic brain injury (TBI) each year in the United States, as many as 75% sustain a mild TBI which can cause long-term or permanent impairments/disabilities in a significant proportion of patients. In addition, traumatic brain injury has become a signature injury of the wars in Iraq and Afghanistan. For people with these injuries, it is difficult to determine whether symptoms are due to the head injury or another condition, such as Post-traumatic Stress Disorder. In this project, there are 3 observational studies that involve testing of mental functions and behavior, imaging of the brain with special x-ray procedures, and blood samples to look at glandular function, which may be affected by head injury. A fourth study is a test of a drug, atorvastatin, which may provide protection for injured brain cells and improve outcome. By collecting and analyzing the information from these tests, it will be possible to make the process of diagnosing mild TBI or post traumatic stress disorder (PTSD) more precise, and also to see if atorvastatin is a helpful drug for patients with MTBI.

DETAILED DESCRIPTION:
Of the more than 1.5 million people who experience a traumatic brain injury (TBI) each year in the United States, as many as 75% sustain a mild TBI (MTBI) which can cause long-term or permanent impairments/disabilities in a significant proportion of patients. In addition, traumatic brain injury has become a signature injury of the wars in Iraq and Afghanistan.

One of the most difficult diagnostic problems is separating the effects of MTBI and post-traumatic stress disorder (PTSD), because signs and symptoms of these conditions often overlap. Early and accurate diagnosis of MTBI and its differentiation from both acute stress disorder (ASD) and PTSD are a major priority for military medicine due to overlap in symptoms (e.g., attention problems) and the frequent lack of external signs or even self-awareness of MTBI, especially in association with blast injury.

The major goals of this project are to improve the ability to diagnose mild traumatic brain injury (MTBI) and to test a drug, atorvastatin, which may improve outcome after MTBI. To accomplish these goals, 200 MTBI subjects and 100 orthopedic injury (OI) subjects, for comparison purposes, will be recruited for variety of clinical evaluations and a phase II drug trial. Only the MTBI subjects will participate in the phase II drug trial, and these subjects may choose to participate only in the observational studies, declining the drug trial.

Potential subjects will be identified in the Emergency Departments (EDs) of two level I trauma centers, located within a few blocks of each other in Houston, Texas. Once discharged from the ED, subjects will be enrolled and baseline procedures will be performed, including behavioral/cognitive testing, sample collection, and medication teaching, including the first dose of study drug. Subjects will be followed by phone at Day 3-4 during the 7-day dosing period of the drug trial, then with return visits for all subjects at one week, one month, three months, and six months after injury.

Investigation of acute civilian MTBI could potentially elucidate the diagnostic issues of distinguishing between MTBI, post-concussion syndrome (PCS), acute stress disorder (ASD), and post-traumatic stress disorder (PTSD) because, in the civilian setting, mild traumatic brain injuries can be characterized prospectively using advanced brain imaging, EEG, and neuropsychological assessment.

We hypothesize that in comparison with OI subjects, the MTBI group will exhibit slowing of EEG frequency, alteration of cerebral white matter microstructure on diffusion tensor imaging (DTI), and cognitive deficit within 24 hours after injury. We also hypothesize that MTBI subjects will show recovery in their EEG frequency and cognition over six months following injury despite residual white matter injury on DTI. We will also collect two plasma samples and a saliva sample, the first within 24 hr of injury (baseline) and the second at six months post-injury, for measurement of potential biomarkers and genetic studies.

Magnetoencephalography (MEG) will be used to detect and characterize focal abnormalities in neurophysiological function in subjects with MTBI diagnosed with PTSD for the purpose of distinguishing between the two. MEG is a completely non-invasive imaging modality which is able to provide information regarding focal abnormalities in the brain. MEG has been shown to be sensitive to cognitive complaints in patients with MTBI and to be more sensitive to these deficits than EEG. In addition, neurophysiological abnormalities found through testing can differentiate patients with MTBI and PTSD in some studies. Thus, we propose to explore the relationship between DTI and MEG findings which may lead to identification of more distinct, replicable patterns of brain abnormalities in subjects with PTSD and MTBI that may lead to better differentiation between these groups of patients and improve diagnostic precision, as well as from patients with a combination of both disorders.

A separate analysis is designed to examine the incidence and effects of hypopituitarism after MTBI. The incidence of hypopituitarism after MTBI is not known. However, in patients who have persistent symptoms at one year post-injury, 35% have been found to have deficiency one or more pituitary hormones. The clinical characteristics, MRI imaging results, EEG and MEG results of the patients who have pituitary deficiency will be compared to those of patients with normal pituitary function. The relationship between pituitary dysfunction and functional outcome, cognitive recovery, and resolution of PCS will be examined as well.

The final component of this protocol is a Phase II randomized clinical trial of the 200 MTBI subjects to evaluate atorvastatin (Lipitor®) as a neuroprotective agent for the treatment of MTBI. The primary endpoint for this trial is three months. This trial will examine the effects of atorvastatin, given orally in a dose of 1mg/kg (up to 80 mg) for seven days, on the development of post-concussive symptoms (PCS), PTSD symptoms, cognitive recovery, and functional outcome at 3 months post-injury, on recovery of EEG and MEG at 3 months post-injury, and on changes in DTI imaging, as well as any effects on liver function.

In conclusion, traumatic brain injury has become the signature injury of the Iraq and Afghanistan wars, and many veterans with mild TBI find their injuries overlooked and misunderstood. The goal of the Mission Connect Mild TBI Translational Research Consortium is to find answers to the challenging questions associated with the diagnosis and treatment of MTBI. The four studies in this Integrated Clinical Protocol begin that process.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years
* MTBI subjects: evidence of closed head injury; Glasgow Coma Score 13-15; loss of consciousness < 30 minutes; post-traumatic amnesia < 24 hours; Abbreviated Injury Score </= 3 for any body region; absence of focal lesions on head CT scan
* Orthopedic Injury subjects: evidence of traumatic injury, other than head; Abbreviated Injury Score </= 3 for any body region
* does not require hospitalization for injuries
* visual acuity and hearing adequate to participate in testing
* fluent in either English or Spanish

Exclusion Criteria:

* Abbreviated Injury Score > 3 for any body region
* any type of penetrating injury
* history of significant pre-existing disease or systemic injuries
* history of schizophrenia or bipolar disorder
* blood alcohol > 200 mL/dL
* left-handed
* existing contraindications for MRI
* claustrophobia
* pregnancy
* exclusions related to atorvastatin, including currently taking any statin drug (atorvastatin, simvastatin, rosuvastatin, pravastatin, lovastatin, fluvastatin), no longer taking a statin drug but history of use within the last six months, previously taking any statin drug at any time but now discontinued due to side effects, taking any medication with known interactions with atorvastatin (cyclosporine, fibric acid derivative, erythromycin, clarithromycin, combination of ritonavir plus saquinavir or lopinavir, niacin in doses exceeding multivitamin dosage, or azole antifungals), active liver disease, history of unexplained persistent elevation of serum transaminases, and hypersensitivity to any component of atorvastatin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia S Robertson, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine/Ben Taub General Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston/Memorial Hermann Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data has been shared through the TED metadataset (https://tbiendpoints.ucsf.edu/ted-metadataset) and plans are to contribute the data to FITBIR as a legacy database.

REFERENCES:
- [Background] King NS, Crawford S, Wenden FJ, Moss NE, Wade DT. The Rivermead Post Concussion Symptoms Questionnaire: a measure of symptoms commonly experienced after head injury and its reliability. J Neurol. 1995 Sep;242(9):587-92. doi: 10.1007/BF00868811. PMID 8551320
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Ware JE Jr., Kosinski M, Turner-Bowker DM, Gandek B. How to Score Version 2 of the SF-12v2® Health Survey [With a Supplement Documenting SF-12® Health Survey] Lincoln, RI: QualityMetric Incorporated, 2002
- [Background] Weathers F, Litz B, Herman D, Huska J, Keane T. The PTSD Checklist [PCL]: Reliability, Validity, and Diagnostic Utility. Paper presented at the Annual Convention of the International Society for Traumatic Stress Studies, San Antonio, TX., October 1993
- [Background] Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. App Psychol Meas. 1977;1:385-401.
- [Derived] Robertson CS, McCarthy JJ, Miller ER, Levin H, McCauley SR, Swank PR. Phase II Clinical Trial of Atorvastatin in Mild Traumatic Brain Injury. J Neurotrauma. 2017 Apr 1;34(7):1394-1401. doi: 10.1089/neu.2016.4717. Epub 2017 Feb 27. PMID 28006970

RESULTS

PARTICIPANT FLOW:
Groups:
- mTBI-atorvastatin Group: 1:1 randomization will be used to assign half of enrolled subjects to the treatment arm. These subjects will receive a daily weight-based dose of atorvastatin 1mg/kg (up to 80 mg) for 7 days starting within 24 hours of mTBI, and their outcome will be compared with the group of subjects receiving a placebo.
- mTBI-placebo Group: 1:1 randomization will be used to assign half of enrolled subjects to the placebo arm. These subjects will receive a daily dose of an inert preparation, visually indistinguishable from the active agent. They will take this preparation for 7 days, starting within 24 hours of mTBI, and their outcome will be compared with the group of subjects receiving atorvastatin.
Period: Overall Study
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Started | 28 | 24
Completed | 27 | 21
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (9.0) | 29.9 (9.9) | 29.5 (9.3)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 20 | 14 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 7 | 18
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Primary Language [Number; unit: participants]
  English | 27 | 21 | 48
  Spanish | 1 | 3 | 4
Education [Number; unit: participants]
  1-8 years | 1 | 1 | 2
  some high school | 1 | 4 | 5
  high school graduate | 8 | 8 | 16
  some college | 12 | 6 | 18
  college graduate | 4 | 3 | 7
  post-graduate | 0 | 1 | 1
  vocational | 2 | 0 | 2
  unknown | 0 | 1 | 1
Galveston Orientation and Amnesia Test Score [Number; unit: participants] — The GOAT assesses the duration of post-traumatic amnesia and was assessed on presentation to the hospital. It includes 10 items on recovery of orientation to person, place, and time and the maximum score is 100. (Levin, H., O'Donnell, V., and Grossman, R. [1979]. The Galveston Orientation and Amnesia Test. A practical scale to assess cognition after head injury. J Nerv Ment Dis 167[11], 675-684.). Categories used were normal (=100) or some abnormality (<100).
  participants
    =100 | 23 | 23 | 46
    <100 | 5 | 1 | 6
Glasgow Coma Scale Score [Number; unit: participants] — GCS was obtained in the emergency room on presentation as an assessment of neurological status. The score has 3 components: eye opening (1-4), verbal response (1-5), and motor response (1-6). The components are summed for a score that ranges from 3-15. Normal GCS is 15, less than 15 indicates some abnormality.
  participants
    15 | 27 | 23 | 50
    14 | 1 | 1 | 2
Head Abbreviated Injury Score [Number; unit: participants] — The head component of the Abbreviated Injury Score describes the severity of a head injury. The score ranges from 1-6, with a higher score indicating a more severe injury. Patients were excluded from this study if any component AIS was greater than 2.
  participants
    1 | 16 | 16 | 32
    2 | 12 | 8 | 20
Injury Severity Score [Mean (Standard Deviation); unit: units on a scale] — ISS is a score that describes the overall injury severity and was determined at presentation to the hospital. There are 9 body regions where the injury severity is assessed on a scale from 1-6, with a higher score indicating a more severe injury. Is all body region scores are < 6, then the ISS is calculated by summing the square of the 3 highest region scores. If any of the body region scores is 6 (unsurvivable) then the ISS is set to 75. The ISS score ranges from 1-75.
  units on a scale | 3.6 (2.0) | 3.5 (1.9) | 3.6 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Rivermead Post-Concussion Symptoms Questionnaire, at 3 Months After Injury.
Description: The Rivermead Post-Concussive Symptoms Questionnaire (RPQ) is a 16-item self-report measure of the presence and severity of the 16 most commonly reported post-concussive symptoms found in the literature. The scale compares any current symptoms to pre-injury symptom levels to account for potential symptom exacerbation due to TBI. The range of scores is 0-64. Values for each of the 16 items include 0 (not experienced at all), 1 (no more of a problem than before the injury), 2 (mild problem), 3 (moderate problem), 4 (severe problem). The total score was a summation of symptoms that represented new symptom onset or an exacerbation of a symptom present pre-injury. (King, N.S., Crawford, S., Wenden, F.J., Moss, N.E., & Wade, D.T. [1995]. The Rivermead Post Concussion Symptoms Questionnaire: A Measure of Symptoms Commonly Experiences after Head Injury and its Reliability. Journal of Neurology 242: 587-92.)
Time Frame: 3 months after injury
Population: The analysis population includes all 27 patients in the atorvastatin group who completed the study and the 21 placebo group patients who completed the study plus one lost to follow-up at 6 months but had completed all of the outcome assessments for the primary and secondary outcomes at 3 months (for a total of 22 placebo group patients).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 2 [0 to 49] | 3.5 [0 to 54]

2. Secondary Outcome: Medical Outcome Study Short Form 12 - Mental Score
Description: SF-12 is a self-report questionnaire that assesses functional health and well-being. There are 12 items in 8 subscales, including physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Physical and Mental Health Composite Scores are computed using the scores of the 12 questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. Both Physical and Mental Health Composite Scales combine the 12 items in such a way that they compare to a national norm with a mean score of 50.0 and a standard deviation of 10.0. (Ware, J.E., Jr., Kosinski, M., Turner-Bowker, D.M., Gandek, B. How to Score Version 2 of the SF-12v2® Health Survey [With a Supplement Documenting SF-12® Health Survey] Lincoln, RI: QualityMetric Incorporated, 2002.)
Time Frame: 3 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 52 [42.75 to 57] | 52 [42.5 to 57.5]

3. Secondary Outcome: Medical Outcome Study Short Form 12 - Physical Score
Description: as for outcome 2
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 55 [51.25 to 57.75] | 56.5 [52 to 58]

4. Secondary Outcome: Post-traumatic Stress Checklist - Civilian Form
Description: The Post Traumatic Stress Disorder Checklist (PCL) is a 17-item self report measure of the DSM-IV symptoms of PTSD. Respondents rate how much they were "bothered by a symptom" on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). The PCL was scored as a total score (range 17-85), with higher total scores indicating more symptoms. (Weathers, F., Litz, B., Herman, D., Huska, J., & Keane, T. [October 1993]. The PTSD Checklist [PCL]: Reliability, Validity, and Diagnostic Utility. Paper presented at the Annual Convention of the International Society for Traumatic Stress Studies, San Antonio, TX.)
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 24 [18 to 29.5] | 21 [19 to 27.25]

5. Secondary Outcome: Connor Davidson Resilience Measure
Description: The Connor-Davidson Resilience scale (CD-RISC) has 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience. The sum score has a range from 0 to 100. (Conner KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale [CD-RISC]. Depress Anxiety 18[2]:76-82,2003].
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 84 [72.25 to 95] | 84 [73.5 to 93]

6. Secondary Outcome: Center for Epidemiological Study Depression Scale
Description: The CES-D is a widely used screening scale for depression, assessing depressive feelings and behaviors occurring in the past week of a patient's life. The CES-D consists of 20 items, which make up six scales reflecting depressive symptomatology: depressed mood, feelings of guilt and worthlessness, feelings of helplessness and hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Each item is scored on a 4-point scale ranging from 0 (rarely/none of the time) to 3 (most/all of the time). Scores for items 4, 8, 12, and 16 are reversed before summing all items to yield a total score, which can range from 0-60. Higher scores indicate more depressive symptoms. (Radloff, LS [1977]. The CES-D Scale: A self-report depression scale for research in the general population. App Psychol Meas, 1, 385-401.)
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 6 [1.25 to 17.0] | 5.5 [3.5 to 11.5]

7. Secondary Outcome: Brief Visuospatial Memory Test - Revised
Description: The BVMT-R is a measure of visuospatial memory. Six equivalent, alternate stimulus forms consist of six geometric figures printed in a 2 x 3 array on separate pages. In three Learning Trials, the subject views the stimulus page for 10 seconds and is asked to draw as many of the figures as possible in their correct location. A Delayed Recall Trial is administered after a 25-minute delay. Last, a Recognition Trial, in which the respondent is asked to identify which of 12 figures were included among the original geometric figures, is administered. Scoring of the immediate and delayed recall are based on the accuracy of the drawings and the location of the figures. For each figure, one point is awarded to each satisfactory domain resulting in a maximum of 12-points per trial.
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 33 [21.25 to 43.5] | 31 [23.3 to 37]

8. Secondary Outcome: Symbol Digit Modalities Test - Oral Score
Description: The SDMT is a measure of divided attention, visual scanning and motor speed. This measure involves a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. The subject is required to scan the key and write down the number corresponding to each symbol as fast as possible. The number of correct substitution within 90 seconds is recorded. In the written version of the test the subject fills in the numbers that correspond to the symbols. In the oral version the examiner records the numbers spoken by the subject. The score is the number of correctly coded items from 0-110 in 90 seconds. A higher score indicates better performance.
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 60 [52 to 70.5] | 68 [53 to 76]

9. Secondary Outcome: Symbol Digit Modalities Test - Written Score
Description: as for outcome 8
Time Frame: 3 months after injury
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Number analyzed (Participants) | 27 | 22
units on a scale | 55 [47.25 to 63] | 55 [45.5 to 66]

ADVERSE EVENTS:
Time Frame: Three months after injury
Arm/Group | mTBI-atorvastatin Group | mTBI-placebo Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/24
Other Adverse Events (participants affected / at risk) | 11/28 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mTBI-atorvastatin Group (N=28) | mTBI-placebo Group (N=24)
constipation (Gastrointestinal disorders) | 4 | 3
abdominal pain (Gastrointestinal disorders) | 1 | 2
fatigue (General disorders) | 3 | 4
fever (General disorders) | 0 | 1
flatulence (Gastrointestinal disorders) | 7 | 6
itching (Skin and subcutaneous tissue disorders) | 1 | 1
diarrhea (Gastrointestinal disorders) | 3 | 2
change in urine (Renal and urinary disorders) | 2 | 1
not feeling well (General disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No